CLINICAL TRIAL: NCT02561611
Title: Multi-component Workplace Energy Balance Intervention
Acronym: WorkACTIVE-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2015-024; R21OH010785-01A1 (NIH)
Record Dates: First submitted 2015-09-23; First posted 2015-09-28 (Estimated); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Obesity
Keywords: Pedal Desk; Workplace Intervention; Physical Activity; Energy Expenditure
MeSH Terms: conditions — Obesity, Abdominal; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): * Usual Working Condition Group (UWC)
  * The no-intervention control condition will be asked to maintain their usual work and lifestyle throughout the study. Participants may be contacted by Pennington Biomedical staff during the intervention.
- Intervention Group (Experimental): * Combined Intervention (Walk More and Pedal Desk; WMPD)
  * Participants in the WMPD condition will engage in both step-counting (Walk More, WM) and pedal desk (PD) intervention components.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — The content of both intervention components will be covered during a weekly scheduled group meeting (or face-to-face meetings, as needed). The step-counting component of the WMPD intervention will be modeled off the success of The First Step Program (FSP).
  Other Names: Walk More and Pedal Desk Group; WMPD
  Arms: Intervention Group

SUMMARY:
The purpose of the WorkACTIVE-P study is to assess the outcome of an innovative multi-component intervention focused on increasing energy expenditure and re-balancing the disrupted energy balance equation of sedentary workplaces with an ultimate target of reducing workers' abdominal obesity.

DETAILED DESCRIPTION:
The energy expenditure intervention includes replacing workplace sedentary time with access to a dedicated pedal desk and increasing steps/day with wearable monitors. Both components are incorporated into an electronically-delivered behavior monitoring and support infrastructure, thus enabling continuous management. The investigators will utilize pedaldesks manufactured and owned by Pennington Biomedical Research Center to conduct this study at Blue Cross Blue Shield of Louisiana offices in Baton Rouge, La. 40 individuals will be recruited and randomized to either a control arm or combined Walk More Pedal Desk (WMPD) intervention. Primary (MRI-determined visceral adipose tissue) and secondary (changes in body weight, total adipose tissue, subcutaneous adipose tissue, blood pressure, blood lipids, fasting glucose and insulin, HbA1-c, free-living accelerometer-determined walking, time spent in sedentary behavior, exercise, and dietary intake) outcomes will be assessed at baseline and month 3.

ELIGIBILITY:
Inclusion Criteria:

* BMI: > or equal to 25.0 kg/m2 and < or equal to 40 kg/m2
* Waist Circumference: >102 cm (men) or > 88 cm (women)
* Any one of the other four defining risk factors defining metabolic syndrome (Triglycerides > or equal to 150 mg/dL , HDL Cholesterol < 40 mg/dL (men) or < 50 mg/dL (women), Resting blood pressure > or equal to 130 mm Hg systolic / 85 mm Hg diastolic, Fasting glucose > or equal to 110 mg/dL)

Exclusion Criteria:

* Systolic blood pressure > 179 mmHg and/or diastolic blood pressure > 99 mmHg
* Self-reported Type 1 or Type 2 diabetes, or use of diabetes-related medications
* Significant CVD or disorders
* Other significant medical conditions including but not limited to implants that may interfere with MRI, chronic respiratory, gastrointestinal, neuromuscular, or psychiatric conditions, malignancies in the past 5 years, with the exception of skin cancer therapeutically controlled, endocrine (including diabetes), any other medical conditions or disease (including arthritis) that is life threatening or that can interfere with or be aggravated by exercise.
* Poor compliance to activity monitors

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorling JL, Hochsmann C, Tudor-Locke C, Beyl R, Martin CK. Effect of an office-based intervention on visceral adipose tissue: the WorkACTIVE-P randomized controlled trial. Appl Physiol Nutr Metab. 2021 Feb;46(2):117-125. doi: 10.1139/apnm-2020-0175. Epub 2021 Jan 15. PMID 33451268

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: * Combined Intervention (Walk More and Pedal Desk; WMPD)
  * Participants in the WMPD condition will engage in both step-counting (Walk More, WM) and pedal desk (PD) intervention components.
  Intervention Group: The content of both intervention components will be covered during a weekly scheduled group meeting (or face-to-face meetings, as needed). The step-counting component of the WMPD intervention will be modeled off the success of The First Step Program (FSP).
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (9.8) | 46.2 (11.4) | 46.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 86.1 (14.0) | 89.6 (16.6) | 87.7 (15.14)

OUTCOME MEASURES:

1. Primary Outcome: Change in Visceral Adipose Tissue (VAT), Measured in kg
Description: Change (end of study minus baseline) in abdominal obesity operationalized as MRI-determined visceral adipose tissue (VAT) and measured in kg.
Time Frame: 3 -month-long controlled trial
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 20 | 20
kg | .04 [-0.07 to 0.15] | -0.10 [-0.22 to 0.01]

2. Secondary Outcome: Changes in Body Weight
Description: Weight will be measured to the nearest 0.1 kg using a standard stadiometer.
Time Frame: 3-month-long controlled trial
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 20 | 20
kg | -0.3 [-1.3 to 0.6] | -0.9 [-1.8 to 0.1]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT02561611/Prot_SAP_000.pdf